CLINICAL TRIAL: NCT02905396
Title: Spinal Cord Stimulation in Small Fibre Neuropathy: A Pilot Study
Brief Title: Spinal Cord Stimulation in Small Fibre Neuropathy
Acronym: SFN-SCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 1 inclusion in 2,5 years
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Catharina G. Faber, Professor, MD, Academisch Ziekenhuis Maastricht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFN-SCS; NL53831.06.15/ METC152054 (Registry Identifier: Medical Ethical Committee Maastricht, the Netherlands)
Record Dates: First submitted 2016-08-23; First posted 2016-09-19 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Small Fiber Neuropathy
Keywords: small fiber neuropathy; spinal cord stimulation; treatment; pain
MeSH Terms: conditions — Small Fiber Neuropathy; Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spinal cord stimulation (Experimental): implantation of spinal cord stimulator
  Interventions: Device: Spinal cord stimulation

INTERVENTIONS:
Device: Spinal cord stimulation — implantation of spinal cord stimulator
  Other Names: Neurostimulation; PrimeAdvanced SureScan MRI-neurostimulator Model 97702 Medtronic

SUMMARY:
Small fibre neuropathy (SFN) is a disorder in which selectively thinly myelinated and unmyelinated nerve fibres are involved. SFN can cause severe and chronic symptoms such as burning pain in the extremities in combination with autonomic symptoms. So far, the results of symptomatic SFN treatment have been rather disappointing, despite the fact that new agents have been developed.

This study is a pilot study to investigate whether Spinal Cord Stimulation (SCS) combined with best (drug) treatment as usual (TAU) leads to clinically significant pain relief in patients suffering from pain in the lower limbs due to SFN, defined as ≥30% pain reduction on a mean NRS during daytime, and/or ≥30% pain reduction on a mean NRS during night-time, and/or at least much improved or very much improved, on the Patient Global Impression of Change (PGIC) for pain and sleep.

DETAILED DESCRIPTION:
Small fibre neuropathy (SFN) is caused by dysfunction of the Aδ-fibres and C-fibres. SFN is diagnosed if there are typical SFN symptoms together with abnormal intraepidermal nerve fibre density (IENFD) in skin biopsy and/or abnormal temperature thresholds in quantitative sensory testing (QST). A large number of disorders can underlie SFN, such as diabetes, amyloidosis, sarcoidosis and other systemic illnesses, vasculitis, and HIV. The proportion of idiopathic or cryptogenic SFN reported in literature varies between 24% and 93%. SFN is not a rare condition; a recent study showed a minimum prevalence of 53/100.000.

SFN can cause severe and chronic symptoms such as burning pain in particularly the extremities in combination with autonomic symptoms, with a significant impact on quality of life. Moreover, neuropathic pain disorders are associated with anxiety, depression and sleep disturbances, polypharmacy and significant healthcare resource use. Therefore, neuropathic pain has a significant impact on society due to the high socioeconomic costs. The treatment of SFN still largely relies on the agents generally used for neuropathic pain relief, particularly derived from diabetic painful neuropathic studies, such as antidepressants (amitriptyline, duloxetine), anti-epileptic agents (pregabalin, gabapentin), opioids and topical agents (lidocain and capsaicin), but have been disappointing in SFN (clinical observation in > 400 patients treated). Therefore it is of major importance to develop new treatment options that can provide sufficient pain relief for the individual patient.

In 1965 Melzack and Wall introduced the gate theory of pain perception. This theory offered new perspectives in treating neuropathic pain. In the seventies SCS was introduced. It was thought that the stimulation of the large myelinated fibres modulates the transmission of pain signals, which run through small, non-myelinated fibres. The exact mechanism of SCS is still unknown. Nowadays SCS is used worldwide and the global sales are estimated for more than 35.000 systems annually. Recently, a prospective two-centre randomized controlled trial was performed to investigate the effect of SCS in painful diabetic polyneuropathy. SCS was successful in 59% of the patients, and the effect lasted for at least 2.5 years in most patients.

The current pilot study will focus on the potential effect of SCS in patients with SFN. The main study parameter will be the mean pain intensity as measured on a Numeric Rating Scale (NRS) and/or a Patient Global Impression of Change (PGIC) for pain and sleep measured on a 7-point Likert scale, after 12 months of treatment in patients with SFN and intractable neuropathic pain in the lower limbs. Besides the primary objective, the following secondary aims are investigated:

1. The effect of SCS on pain (at least 30% pain reduction, on mean daily, night, and maximum pain);
2. the effect of SCS on activity and participation;
3. the effect of SCS on and health related quality of life;
4. the effect of SCS on mood in SFN;
5. the effect of SCS on the reduction of pain medication.

ELIGIBILITY:
Inclusion Criteria:

* SFN diagnosis according to international criteria,
* Age between 18 and 75 years, lucid,
* Mean pain intensity during daytime or night-time should be 5 or higher on the 11-points numeric rating scale (NRS),
* The pain intended to treat has been present for more than 12 months, as declared by patients to the best of their knowledge or after studying available medical records,
* Previous treatment has been unsuccessful (insufficient pain relief and/or unacceptable side-effects) with drugs from the following drug categories

  * Tricyclic anti-depressant agent (e.g., Amitriptyline)
  * Alpha 2-delta calcium channel agonist/Anti-epileptic drugs (e.g. Pregabalin (Lyrica) or Gabapentin (Neurontin)),
  * Serotonin-norepinephrine reuptake inhibitors (e.g., Duloxetine (Cymbalta)),
  * Tramadol or strong opioids.
* Patients will have to be treated or have been treated with at least 3 drugs from the above mentioned drug categories according to the EFNS guidelines for neuropathic pain [34]. Starting dosage is based on individual patient characteristics. Each drug has to be tried for at least 3 weeks and dose will have to be raised once, if possible. Drug treatment can be stopped due to insufficient pain relief and/or unacceptable adverse events.
* Patients will have to be in steady state in medication use for at least 2 months prior to inclusion.

Exclusion Criteria:

* Neuromodulation in history,
* Neuropathic pain prevalent in the upper limbs (UL) compared to the legs; UL NRS not exceeding 3)
* Neuropathy or chronic pain of other origin than SFN (NRS > 3),
* Addiction: drugs, alcohol (5E / day) and/or specific medication

  * Drugs: cocaine, heroin, marihuana,
  * Alcohol: wine, beer, liquor,
  * Medication: benzodiazepines.
* Insufficient cooperation from the patient (little motivation, understanding or communication problems),
* Blood clotting disorder or the use of oral anticoagulation that cannot be stopped for a period of 10 days around the implantation procedure.
* Immune deficiency (HIV-positive if known, corticosteroids with a dose equivalent to > prednisolone 10 mg, immunosuppressive medication, etc.)
* Known peripheral vascular disease, no palpable peripheral pulsations at the feet (inclusion is possible if pulsations are absent, but ankle/brachial index is between 0.7 and 1.2 in both feet)
* Life expectancy < 1 year
* Pacemaker
* Local infection or other skin disorders at site of incision
* Other clinically significant or unstable, or severe acute or chronic medical or psychiatric/psychological condition or laboratory abnormality that may increase the risk associated with study participation or procedure or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Pregnancy
* Severe cardiac or pulmonary failure (> NYHA classification II)
* Use of opioids (higher dose than an equivalent of 30 mg morphine a day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Pain relief | Up to 1 year
  The primary objective of this study is to investigate whether SCS combined with best (drug) treatment as usual (TAU) leads to clinically significant (≥30%) pain relief in patients suffering from pain in the lower limbs due to SFN after 12 months of treatment.
  Clinical significant pain relief is determined as:
  1. ≥30% pain reduction on the mean daytime pain using the NRS, and/or
  2. ≥30% pain reduction on the night-time pain using the NRS and/or
  3. At least much improved or very much improved on the Patient Global Impression of Change (PGIC) for pain and sleep.

SECONDARY OUTCOMES:
Pain reduction | Up to 1 year
  The effect of SCS on pain. Number of patient with a pain reduction of ≥50% on a mean daytime, night-time and maximum pain (separately examined) using the PI-NRS.
Activity and participation | Up to 1 year
  The effect of SCS on activity and participation: questionnaire
Quality of life | Up to 1 year
  The effect of SCS on health related QoL in SFN: questionnaire
Mood | Up to 1 year
  The effect of SCS on mood in SFN: questionnaire
Reduction of pain medication | Up to 1 year
  The effect of SCS on the reduction of pain medication: questionnaire
Change in SFN symptoms | Up to 1 year
  The effect of SCS on a change in SFN symptoms will be measured by the symptom inventory questionnaire (SFN-SIQ) at baseline, 2 weeks, 3, 6, 9, and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands